CLINICAL TRIAL: NCT06551285
Title: Study of the Effect of a Nutritional Supplement on Microbiota, Metabolic Control, Inflammatory Profile, and Quality of Life in Patients With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celia Bañuls (Other)
Responsible Party: Sponsor-Investigator, Celia Bañuls, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIm: 131/23
Record Dates: First submitted 2024-07-31; First posted 2024-08-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Syndrome
Keywords: Insulin resistance; Inflammation; Oxidative Stress; Intestinal microbiota
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary supplement in PCOS (Active Comparator): Subjects will recieve nutritional intervention by a registered dietitian and a supplement containing inositol, vitamin D, zinc, and curcumin for 3 months. The dietary intervention consists of healthy dietary recommendations and hipocaloric diet if needed (overweight, obesity).
  Interventions: Dietary Supplement: Ovapro (Lifepro)
- Placebo in PCOS (Placebo Comparator): Subjects will recieve nutritional intervention by a registered dietitian and a supplement containing yellow colorant for 3 months. The dietary intervention consists of healthy dietary recommendations and hipocaloric diet if needed (overweight, obesity).
  Interventions: Dietary Supplement: Ovapro (Lifepro)
- No intervention in healthy subjects (No Intervention): Healthy subjects will not recieve supplement/placebo nor dietary intervention.

INTERVENTIONS:
Dietary Supplement: Ovapro (Lifepro) — Dietary supplement that contains inositol, vitamin D, zinc, and curcumin.
  Arms: Dietary supplement in PCOS; Placebo in PCOS

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a complex endocrine-metabolic disorder characterized by elevated androgen levels due to ovarian overproduction. Although the pathophysiology of PCOS is not fully understood, it is estimated that insulin resistance (IR) occurs in 70-80% of PCOS cases, which may contribute to hyperandrogenism in affected women.

Women with PCOS and IR are more likely to develop metabolic syndrome, increasing the risk of diabetes, cardiovascular diseases, lipid profile deterioration, elevated inflammation levels, and greater oxidative stress.

The symptoms of PCOS are varied and differ among patients. Common symptoms include androgenic alopecia, hirsutism, acne, abdominal fat accumulation, and fertility issues. These physical manifestations and related problems have been associated with reduced quality of life and self-esteem in these women. The symptoms of PCOS can be improved through lifestyle changes aimed at enhancing insulin sensitivity, such as proper nutrition and regular physical exercise.

Some supplements, such as a combination of Myo-inositol and D-chiro-inositol in a 40:1 ratio, are being used to support the management of PCOS because they appear to improve insulin sensitivity, as well as reduce underlying inflammation and oxidative stress.

To determine whether nutritional intervention combined with inositol supplementation improves PCOS symptoms, various variables will be analyzed to assess improvements in oxidative stress markers, inflammation, lipid profile, hormonal profile, and microbiota. Additionally, if the metabolic profile improves, it is hypothesized that this could also enhance quality of life and self-esteem.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is an endocrine-metabolic disorder that affects many women of reproductive age. PCOS is not just a reproductive disorder but a systemic condition, as cases of PCOS have been described even in menopause, although its prevalence in post-reproductive stages is not high. The diagnosis of PCOS is made using the Rotterdam criteria, agreed upon in 2003 by ESHRE and ASRM (European Society for Human Reproduction and Embryology/American Society for Reproductive Medicine). According to these criteria, a patient must meet two of the following three criteria to be diagnosed with PCOS: oligo-anovulation, clinical or biochemical hyperandrogenism, and polycystic ovarian appearance.

The Rotterdam criteria are widely used but can sometimes lead to an erroneous diagnosis of PCOS. Therefore, in 2006, the AES (Androgen Excess Society) decided that, in addition to the 2003 Rotterdam criteria, hyperandrogenism-either physical or biochemical-was necessary for a PCOS diagnosis. Depending on the criteria used and the diversity of the population studied, epidemiological results can vary. Despite this variability, it is estimated that PCOS affects 6-12% of women of reproductive age.

The most common manifestations of PCOS include androgenic alopecia, hirsutism, acne, irregular cycles, or periods of amenorrhea. An ultrasound image showing polycystic ovarian morphology alone is insufficient for diagnosing PCOS. In polycystic ovaries, more than 12 follicles of 2-9 mm in size and increased ovarian volume (>10 ml) should be visualized using transvaginal ultrasound. Despite the complex and not fully understood pathophysiology of PCOS, two main types of alterations are identified.** On one hand, there is an accelerated release of gonadotropin-releasing hormone (GnRH), which leads to an increased release of luteinizing hormone (LH), resulting in greater androgen production, altered folliculogenesis, and long menstrual cycles or amenorrhea. On the other hand, there is an alteration in ovarian steroidogenesis and folliculogenesis due to increased activity of cytochrome P450c17, an enzyme involved in the synthesis of ovarian and adrenal androgens, leading to elevated androgen levels.

In 70-80% of PCOS cases, women present insulin resistance (IR), with 30-50% of these also exhibiting obesity. High body fat percentage and hyperinsulinemia play significant roles in the development and progression of PCOS. Chronically elevated insulin levels can be associated with elevated androgen levels in a bidirectional manner. Elevated insulin levels may stimulate LH production and increase the activity of the P450c17 enzyme in the ovaries and adrenal glands, resulting in reduced hepatic production of sex hormone-binding globulin (SHBG), which increases the amount of free androgens. Conversely, elevated androgens are associated with increased insulin resistance in the muscles, leading to poorer glucose uptake.

Obesity is considered an amplifying factor in the pathophysiology of PCOS. Adipose tissue is an endocrine organ, and a high amount of adipose tissue increases the production of inflammatory cytokines, which can worsen IR by interfering with glucose uptake. While 70-80% of women with PCOS have IR, there is a 20-30% subgroup without metabolic involvement. Women with PCOS who have a healthy body fat percentage also present with insulin resistance, suggesting that obesity is not the cause of PCOS.

PCOS is a syndrome with a significant genetic basis, complex, and multifactorial pathophysiology. Lifestyle benefits in improving symptoms and the syndrome's progression are an important therapeutic tool. PCOS directly affects the quality of life of patients due to the long-term symptoms and comorbidities associated with this condition, such as obesity, type 2 diabetes mellitus (T2DM), metabolic syndrome (MS), and psychological and emotional issues. Consequently, women with PCOS generally have poorer health compared to those without the condition. Furthermore, comorbidities directly impact quality of life and individual perception of it.

To improve symptoms and prevent the comorbidities, the first line of treatment for patients with PCOS and IR should involve lifestyle modifications. Nutritional intervention and physical exercise are fundamental in maintaining a proper body composition, which can prevent the worsening of PCOS symptoms. The quality and composition of the diet are crucial, beyond the implications of body weight. A hypocaloric diet including low glycemic load foods has been shown to improve the homeostatic model assessment of insulin resistance (HOMA-IR), low-density lipoprotein (LDL) levels, triglycerides (TGC), cholesterol, and free androgen index (FAI). Improving lifestyle will directly impact body fat percentage, which, in turn, will improve hyperandrogenism and ovarian function.

Mental health disorders are highly prevalent among women with PCOS, particularly anxiety, depression, and sleep disorders. Sleep disturbances impact the onset and progression of anxiety and depression in PCOS patients; thus, treating sleep-related issues should be part of the overall treatment. Sleep deprivation is associated with an increased risk of IR, obesity, and type 2 diabetes (T2D). It has been observed that patients with PCOS have decreased melatonin levels in follicular fluid. Melatonin is a potent antioxidant that protects ovarian follicles during maturation. Therefore, sleep disorders can worsen insulin resistance and consequently exacerbate PCOS with metabolic involvement.

Additionally, the microbiota, through the production of various metabolites, impacts complex mechanisms such as hunger and satiety regulation, carbohydrate and lipid metabolism, which can directly affect body composition and PCOS symptoms. The gut microbiota can regulate up to 10% of the transcriptome and host genes involved in metabolism, proliferation, and immune response. Moreover, diet can modulate the gut microbiota composition in patients with PCOS and IR, as an increase in bifidobacteria correlates with improved insulin sensitivity and reduced inflammation. Short-chain fatty acids (SCFAs) such as acetate and butyrate, produced by beneficial gut microbiota, influence glycemia. Given the role of these metabolites in carbohydrate and lipid metabolism, achieving a healthy microbiota state could be a therapeutic goal to reduce systemic inflammation and improve IR.

The two specific inositol stereoisomers, Myo-inositol (MI) and D-chiro-inositol (DCI), act as second messengers of insulin. MI transforms into an insulin second messenger, Myo-inositol phosphoglycan (MI-IPG), which is involved in cellular glucose uptake, while DCI converts into another insulin second messenger, DCI-IPG, which is involved in glycogen synthesis. In patients with PCOS, there appears to be an increased epimerization of Myo-inositol (MI) to D-chiro-inositol (DCI) at the ovarian level due to insulin's effect. Consequently, there is an excess of DCI and a deficiency of MI, which can affect follicle-stimulating hormone (FSH) signaling and deteriorate oocyte quality. Therefore, inositol supplementation is considered an effective and safe method for improving PCOS symptoms by enhancing insulin sensitivity, follicular development, and oocyte maturation. This insulin-sensitizing effect of inositol can help normalize blood androgen levels and improve glycemia. Metformin is a common treatment for women with PCOS and IR. Recent results show that Myo-inositol can be as effective as metformin without its side effects. Both inositol and metformin can improve the metabolic and clinical profile of PCOS patients, as well as metabolic disorders related to diabetes.

Additionally, adequate vitamin D levels should also be considered in patients with PCOS, as vitamin D is involved in increasing the synthesis and release of insulin, enhances insulin receptor presence, and improves insulin response in glucose transport. Vitamin D indirectly affects carbohydrate metabolism by normalizing extracellular calcium levels and parathyroid hormone concentration. It also impacts systemic inflammation by inhibiting the production of pro-inflammatory cytokines, which could contribute to the development of IR. Patients with PCOS who took 20,000 IU of cholecalciferol (Vitamin D) weekly benefited from improved carbohydrate metabolism and better menstrual frequency. Combined supplementation of magnesium, zinc, calcium, and vitamin D in another study led to a significant reduction in total testosterone compared to placebo, although it did not affect sex hormone-binding globulin (SHBG) levels or the free androgen index (FAI). However, the combination of vitamin D and fish oil reduced inflammation markers in the body, such as serum C-reactive protein (CRP), downregulated interleukin 1 (IL-1), and total testosterone levels. A beneficial effect on mental health parameters was also observed, assessed through the Beck Depression Inventory. Available literature shows that zinc supplementation may be indicated in patients with PCOS, as zinc plays an important role in glucose and lipid metabolism. Zinc deficiency may play a significant role in PCOS pathophysiology and also serve as a prognostic marker for the syndrome. It appears that zinc levels in PCOS patients are significantly lower compared to healthy controls. Low zinc intake in individuals with high body fat percentage is associated with hyperinsulinemia, low-grade inflammation, and deterioration of the lipid profile. Zinc ions can act as insulin mimetics in adipocytes, stimulating lipogenesis and glucose transport through the translocation of glucose transporter 4 (GLUT4) to the plasma membrane.

In PCOS patients, there is known to be higher oxidative stress, which could worsen the symptoms of PCOS. Curcumin, extracted from turmeric (Curcuma longa), is a biologically active phytochemical with antioxidant properties. Studies with curcumin in animals have shown promising results, but in PCOS patients, the literature is inconclusive, and it is limited to suggesting that curcumin may have beneficial effects in the clinical management of PCOS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45 years.
* Patients diagnosed with PCOS using the AE-PCOS diagnostic criteria (2009).
* Patients who agree to participate in the study and sign the informed consent form after reading it.

Exclusion Criteria:

* Having been treated with medication or supplementation aimed at improving PCOS prior to the study (e.g., metformin, hormonal therapy, inositol, etc.).
* Suffering from an infectious, hematological, inflammatory, or autoimmune disease.
* Having a severe organic disease.
* Suffering from cardiovascular disease (heart attack, ischemia, thromboembolism).
* Diabetes Mellitus.
* Severe arterial hypertension.
* Alcoholism.
* Active smoking.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological female gender.
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Verify that nutritional intervention and inositol supplementation improve the symptoms of PCOS. | 5 years
  To assess if there is an improvement in PCOS symptoms, both PCOSQ and Ferriman-Gallwey test and regularity of menstrual cycle will be evaluated.
  PCOSQ result must be assessed as 7-point scales in which 7 represents optimal function and 1 represents the poorest function.
  Ferriman-Gallway test gives a total score, which can range from 0 to 36. A score of ≥8 si considered a sign of androgen excess in caucausian women; a score of 8-15 indicates mild hirsutism, and >15 indicates moderate or severe hirsutism.
  The classification of patients between PCOS or healthy will be carried out using Rotterdam criteria.
Evaluate the differences in the diversity of the intestinal microbiota depending on whether patients present PCOS or not. | 5 years
  To asses the differences in alpha-diversity of the intestinal microbiota in both groups, it will be evaluated whether there are significant differences between the Shannon indices of the two groups.

SECONDARY OUTCOMES:
Evaluate significant changes in body fat mass percentage after the dietetic intervention and dietetic supplement. | 3 years
  Percentage of body fat mass will be measured by bioelectrical impedance. It is considered to be high when ≥30% in women. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in high-sensitivity C-reactive protein (hs-CRP) as an inflammatory parameter after the dietary intervention and dietetic supplement. | 3 years
  Participants will be considered to have achieved an improvement in high-sensitivity C-reactive protein levels if they normalize its value (normality values defined between 0 and 1.69mg/dl).
Evaluate significant changes in C3 protein as an inflammatory parameter after the dietetic intervention and dietetic supplement. | 3 years
  Participants will be considered to have achieved an improvement in C3 protein if they normalize its value (normality values defined between 81 and 157mg/dl).
Evaluate significant changes in interleukin 1-beta (IL-1B) levels as a pro-inflammatory molecule after the dietetic intervention and dietetic supplement. | 3 years
  IL-1B levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in interleukin 6 (IL-6) levels as a pro-inflammatory molecule after the dietetic intervention and dietetic supplement. | 3 years
  IL-6 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in tumor necrosis factor alpha (TNF-alpha) levels as a pro-inflammatory molecule after the dietetic intervention and dietetic supplement. | 3 years
  TNF-alpha levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in superoxide dismutase (SOD) levels after the dietetic intervention and dietetic supplement. | 3 years
  Superoxide dismutase levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate if there is a significant reduction after the dietetic intervention in total ROS levels. | 3 years
  Total ROS levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess if there is a significant reduction after the dietetic intervention in glutathione levels. | 3 years
  Total glutathione levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant change after the dietetic intervention in total free radicals and superoxide levels. | 3 years
  Total free radicals and superoxide content will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant reduction after the dietetic intervention in mitochondrial ROS production. | 3 years
  Mitochondrial ROS production will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate if there is a significant improvement after the dietetic intervention in mitochondrial membrane potential. | 3 years
  Mitochondrial membrane potential will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sander VA, Hapon MB, Sicaro L, Lombardi EP, Jahn GA, Motta AB. Alterations of folliculogenesis in women with polycystic ovary syndrome. J Steroid Biochem Mol Biol. 2011 Mar;124(1-2):58-64. doi: 10.1016/j.jsbmb.2011.01.008. Epub 2011 Jan 22. PMID 21262361
- [Background] Sachdeva G, Gainder S, Suri V, Sachdeva N, Chopra S. Obese and Non-obese Polycystic Ovarian Syndrome: Comparison of Clinical, Metabolic, Hormonal Parameters, and their Differential Response to Clomiphene. Indian J Endocrinol Metab. 2019 Mar-Apr;23(2):257-262. doi: 10.4103/ijem.IJEM_637_18. PMID 31161114
- [Background] Panidis D, Tziomalos K, Misichronis G, Papadakis E, Betsas G, Katsikis I, Macut D. Insulin resistance and endocrine characteristics of the different phenotypes of polycystic ovary syndrome: a prospective study. Hum Reprod. 2012 Feb;27(2):541-9. doi: 10.1093/humrep/der418. Epub 2011 Dec 5. PMID 22144419
- [Background] Navarro G, Allard C, Xu W, Mauvais-Jarvis F. The role of androgens in metabolism, obesity, and diabetes in males and females. Obesity (Silver Spring). 2015 Apr;23(4):713-9. doi: 10.1002/oby.21033. Epub 2015 Mar 6. PMID 25755205
- [Background] Jamil AS, Alalaf SK, Al-Tawil NG, Al-Shawaf T. A case-control observational study of insulin resistance and metabolic syndrome among the four phenotypes of polycystic ovary syndrome based on Rotterdam criteria. Reprod Health. 2015 Jan 16;12:7. doi: 10.1186/1742-4755-12-7. PMID 25595199
- [Background] Toosy S, Sodi R, Pappachan JM. Lean polycystic ovary syndrome (PCOS): an evidence-based practical approach. J Diabetes Metab Disord. 2018 Nov 13;17(2):277-285. doi: 10.1007/s40200-018-0371-5. eCollection 2018 Dec. PMID 30918863
- [Background] Szczuko M, Skowronek M, Zapalowska-Chwyc M, Starczewski A. Quantitative assessment of nutrition in patients with polycystic ovary syndrome (PCOS). Rocz Panstw Zakl Hig. 2016;67(4):419-426. PMID 27925712
- [Background] Yang Y, Deng H, Li T, Xia M, Liu C, Bu XQ, Li H, Fu LJ, Zhong ZH. The mental health of Chinese women with polycystic ovary syndrome is related to sleep disorders, not disease status. J Affect Disord. 2021 Mar 1;282:51-57. doi: 10.1016/j.jad.2020.12.084. Epub 2020 Dec 27. PMID 33388474
- [Background] Mojaverrostami S, Asghari N, Khamisabadi M, Heidari Khoei H. The role of melatonin in polycystic ovary syndrome: A review. Int J Reprod Biomed. 2019 Dec 30;17(12):865-882. doi: 10.18502/ijrm.v17i12.5789. eCollection 2019 Dec. PMID 31970309
- [Background] Jiao N, Baker SS, Nugent CA, Tsompana M, Cai L, Wang Y, Buck MJ, Genco RJ, Baker RD, Zhu R, Zhu L. Gut microbiome may contribute to insulin resistance and systemic inflammation in obese rodents: a meta-analysis. Physiol Genomics. 2018 Apr 1;50(4):244-254. doi: 10.1152/physiolgenomics.00114.2017. Epub 2018 Jan 26. PMID 29373083
- [Background] Zhang Z, Bai L, Guan M, Zhou X, Liang X, Lv Y, Yi H, Zhou H, Liu T, Gong P, Sun J, Zhang L. Potential probiotics Lactobacillus casei K11 combined with plant extracts reduce markers of type 2 diabetes mellitus in mice. J Appl Microbiol. 2021 Oct;131(4):1970-1982. doi: 10.1111/jam.15061. Epub 2021 Apr 8. PMID 33694236
- [Background] Bamberger C, Rossmeier A, Lechner K, Wu L, Waldmann E, Fischer S, Stark RG, Altenhofer J, Henze K, Parhofer KG. A Walnut-Enriched Diet Affects Gut Microbiome in Healthy Caucasian Subjects: A Randomized, Controlled Trial. Nutrients. 2018 Feb 22;10(2):244. doi: 10.3390/nu10020244. PMID 29470389
- [Background] den Besten G, van Eunen K, Groen AK, Venema K, Reijngoud DJ, Bakker BM. The role of short-chain fatty acids in the interplay between diet, gut microbiota, and host energy metabolism. J Lipid Res. 2013 Sep;54(9):2325-40. doi: 10.1194/jlr.R036012. Epub 2013 Jul 2. PMID 23821742
- [Background] Heimann E, Nyman M, Palbrink AK, Lindkvist-Petersson K, Degerman E. Branched short-chain fatty acids modulate glucose and lipid metabolism in primary adipocytes. Adipocyte. 2016 Oct 28;5(4):359-368. doi: 10.1080/21623945.2016.1252011. eCollection 2016 Oct-Dec. PMID 27994949